CLINICAL TRIAL: NCT02486380
Title: Toffee Full Face and Toffee Nasal Mask Evaluation in Obesity Hypoventilation Syndrome (NZ)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment terminated permanently due to limited resource to recruit.
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-162
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Full face/Nasal masks (Experimental): Toffee Full face/Toffee nasal
  Interventions: Device: Toffee full face mask/toffee nasal mask

INTERVENTIONS:
Device: Toffee full face mask/toffee nasal mask — Toffee full face mask/toffee nasal mask

SUMMARY:
This investigation is to evaluate the performance, comfort and ease of use of the Toffee full face and toffee nasal mask masks amongst Obesity Hypoventilation Syndrome (OHS) patients in an overnight study.

DETAILED DESCRIPTION:
Up to 20 OHS patients who currently use a full face mask or a nasal mask will be recruited. They will be issued a F&P Toffee Full face (if they are existing full face users) or F&P Toffee Nasal (if they are existing nasal users) for an overnight polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* Diagnosed with OHS by a practicing physician
* Existing full face mask user or a nasal mask user
* Prescribed PAP therapy (Bi-Level or CPAP)

Exclusion Criteria:

* Inability to give informed consent
* Pregnant or think they may be pregnant
* Anatomical or physiological conditions making PAP therapy inappropriate
* Patients requiring supplemental oxygen with their PAP device
* Patients who are in a coma or decreased level of consciousness
* Existing Toffee full face and Toffee nasal mask users
* No arterial PCO2 value from their medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Objective Leak data | 1 night
  Obtained from the participant's device and polysomnography (PSG)

SECONDARY OUTCOMES:
Subjective measurement of Leak | 1 night
  Questionnaire
Comfort | 1 night
  Questionnaire
Ease of use | 1 night
  Questionnaire
Sleep efficiency | 1 night
  Obtained through the PSG
Wake after Sleep Onset (WASO) | 1 night
  Obtained through the PSG
Arousal Index (AI) | 1 night
  Obtained through the PSG

CONTACTS AND LOCATIONS:
Overall Officials: Bhavi Ogra, BSc, Principal Investigator — Fisher & Paykel Healthcare
Locations (1):
- Fisher & Paykel Healthcare, Auckland, New Zealand